CLINICAL TRIAL: NCT04046796
Title: Genetic Causes of Discrepant Clinic in Monogenic Twins
Acronym: DISCO-TWIN
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: DISCO-TWIN
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rare Diseases; Genetic Predisposition to Disease
Keywords: Rare Diseases; Genetic Predisposition; Omics Technology; Next Generation Sequencing (NGS)
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling for NGS analysis and other omics analysis (transcriptomics, proteomics, metabolomics), functional cell biology studies (for example in fibroblast cultures).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy twin
  Interventions: Genetic: NGS Diagnostic
- Effected Twin: Twin with unclear rare diseases, clinically characterized in the context of outpatient/ inpatient standard care at the University Hospital Tübingen (UKT) or cooperating location.
  Interventions: Genetic: NGS Diagnostic

INTERVENTIONS:
Genetic: NGS Diagnostic — Blood take for genetic diagnostic.
  Other Names: Omics Technology

SUMMARY:
In the DISCO-TWIN study (prospective, open-label molecular-genetic study), twin pairs with one healthy and one affected twin with molecularly undiagnosed diseases will be analysed by means of omics technologies and/ or re-analysed using existing datasets. Phenotype and omics data will be shared within the University Hospital Tübingen and with external collaborators to improve the diagnostic rate of the subjects included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Twin pair monozygotic clinically (phenotypic) discordant twins
* Unclear diagnosis
* Suspected (mono-)genetic cause of the disease in one twin

Exclusion Criteria:

* Missing informed consent of both twin/ legal representative
* No distinct phenotype

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twin pair monozygotic clinically (phenotypic) discordant twins
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of new Candidate Genes | Day 1
  Number of new Candidate Genes for complex or serious diseases through a comparative genetic analysis of monozygotic clinically discordant twins

SECONDARY OUTCOMES:
Number of putative disease causes | Day 1
  Number characterizations of the identified putative disease causes.
Number of diagnosis | Day 1
  Number of patients receiving appropriate therapy after successful diagnosis
Number of molecular causes of diagnostically unclear rare diseases | Day 1
  Number of molecular causes of diagnostically unclear rare diseases

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Hübener-Schmid, Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No